CLINICAL TRIAL: NCT00077636
Title: A Randomized, Open-label Study of the Effect of PEGASYS and Ribavirin Combination Therapy on Sustained Virologic Response in Interferon-naïve Patients With Chronic Hepatitis C Genotype 2 or 3 Infection
Brief Title: ACCELERATE Study - A Study of PEGASYS (Peginterferon Alfa-2a (40KD)) in Combination With COPEGUS (Ribavirin) in Interferon-Naive Patients With Chronic Hepatitis C (CHC) Infection.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NV17317
Record Dates: First submitted 2004-02-10; First posted 2004-02-13 (Estimated); Results first posted 2016-01-21 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-01

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Copegus; Drug: peginterferon alfa-2a [Pegasys]
- 2 (Experimental)
  Interventions: Drug: Copegus; Drug: peginterferon alfa-2a [Pegasys]

INTERVENTIONS:
Drug: Copegus — 400mg po bid for 16 weeks
  Arms: 1
Drug: Copegus — 400mg po bid for 24 weeks
  Arms: 2
Drug: peginterferon alfa-2a [Pegasys] — 180 micrograms sc weekly for 16 weeks
  Arms: 1
Drug: peginterferon alfa-2a [Pegasys] — 180 micrograms sc weekly for 24 weeks
  Arms: 2

SUMMARY:
This study will evaluate the efficacy and safety of different durations of treatment with PEGASYS combined with ribavirin in patients with CHC genotype 2 or 3 infection who have never previously received interferon (IFN) therapy. The anticipated time on study treatment is 3-12 months and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* patients >=18 years of age;
* CHC infection (genotype 2 or 3);
* liver biopsy (in <24 calendar months of first dose), with results consistent with CHC infection;
* use of 2 forms of contraception during study and 6 months after the study in both men and women.

Exclusion Criteria:

* women who are pregnant or breastfeeding;
* male partners of women who are pregnant;
* conditions associated with decompensated liver disease;
* other forms of liver disease, including liver cancer;
* human immunodeficiency virus infection;
* previous treatment with an IFN, pegylated IFN, ribavirin, viramidine, levovirin, or amantadine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1469 (Actual)
Dates: Start 2003-12; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (117):
- United States (78):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Anchorage, Alaska
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Little Rock, Arkansas
  - La Jolla, California
  - Long Beach, California
  - Los Angeles, California
  - Palo Alto, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - San Luis Obispo, California
  - Littleton, Colorado
  - Farmington, Connecticut
  - Bradenton, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Tampa, Florida
  - Wellington, Florida
  - Atlanta, Georgia
  - Austell, Georgia
  - Honolulu, Hawaii
  - Boise, Idaho
  - Moline, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Baton Rouge, Louisiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Plymouth, Minnesota
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - Bayside, New York
  - Binghamton, New York
  - Manhasset, New York
  - New York, New York
  - The Bronx, New York
  - Williamsville, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Fayetteville, North Carolina
  - Statesville, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Lancaster, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Cranston, Rhode Island
  - Providence, Rhode Island
  - Germantown, Tennessee
  - Dallas, Texas
  - Fort Sam Houston, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - White River Junction, Vermont
  - Charlottesville, Virginia
  - Chesapeake, Virginia
  - Falls Church, Virginia
  - Richmond, Virginia
  - Bellevue, Washington
  - Kirkland, Washington
  - Puyallup, Washington
  - Seattle, Washington
  - Spokane, Washington
  - Madison, Wisconsin
  - Cheyenne, Wyoming
- Australia (5):
  - Adelaide
  - Brisbane
  - Kingswood
  - Melbourne
  - Woolloongabba
- Canada (3):
  - Edmonton, Alberta
  - Downsview, Ontario
  - Mississauga, Ontario
- France (9):
  - Clichy
  - Créteil
  - La Tronche
  - Marseille
  - Nice
  - Rennes
  - Strasbourg
  - Toulouse
  - Vandœuvre-lès-Nancy
- Germany (6):
  - Berlin
  - Düsseldorf
  - Freiburg im Breisgau
  - Hanover
  - Homburg/saar
  - Kiel
- Italy (6):
  - Bergamo
  - Bologna
  - Milan
  - Napoli
  - Pavia
  - Pisa
- Otahuhu, New Zealand
- Puerto Rico (3):
  - Ponce
  - San Juan
  - Santurce
- Spain (6):
  - Badalona
  - Barakaldo
  - Barcelona
  - Madrid
  - Seville
  - Valencia

REFERENCES:
- [Derived] Shiffman ML, Suter F, Bacon BR, Nelson D, Harley H, Sola R, Shafran SD, Barange K, Lin A, Soman A, Zeuzem S; ACCELERATE Investigators. Peginterferon alfa-2a and ribavirin for 16 or 24 weeks in HCV genotype 2 or 3. N Engl J Med. 2007 Jul 12;357(2):124-34. doi: 10.1056/NEJMoa066403. PMID 17625124

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 8 countries from 20 November 2003 to 13 September 2005.
Pre-assignment Details: A total of 1400 participants were planned for the study; 1469 were randomized (736 were assigned to the 16-week treatment group and 733 were assigned to the 24-week treatment group) and 1465 received the study treatment.
Groups:
- PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 16 Weeks: Participants received 180 micrograms (mcg) of PEG-IFN alfa-2a once weekly and 800 milligrams (mg) of ribavirin daily for 16 weeks.
- PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 24 Weeks: Participants received 180 mcg of PEG-IFN alfa-2a once weekly and 800 mg of ribavirin daily for 24 weeks.
Period: Overall Study
Arm/Group | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 16 Weeks | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 24 Weeks
Started | 736 | 733
Completed | 692 | 641
Not Completed | 44 | 92
Not completed — Refused Treatment | 9 | 31
Not completed — Admin | 3 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Adverse Event | 17 | 34
Not completed — Protocol Violation | 0 | 2
Not completed — Lost to Follow-up | 10 | 18
Not completed — Abnormality Of Laboratory Test | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 16 Weeks: Participants were administered 180 micrograms (μg) of PEG-IFN alfa-2a once weekly and 800 milligrams (mg) of ribavirin daily for 16 weeks.
- PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 24 Weeks: Participants were administered 180 μg of PEG-IFN alfa-2a once weekly and 800 mg of ribavirin daily for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 16 Weeks | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 24 Weeks | Total
Number analyzed (Participants) | 736 | 733 | 1469
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.1 (9.83) | 45.6 (9.98) | 45.8 (9.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 285 | 271 | 556
  Male | 451 | 462 | 913

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virological Response (SVR)
Description: SVR was defined as the percentage of participants with undetectable HCV RNA at 24 weeks after the completion of the study treatment. The negative assessment was required to be the last one collected at or after week 36 (ie, on or after study Day 253) for the 16-week treatment group or at or after week 44 (ie, on or after study Day 309) for the 24-week treatment group.
Time Frame: Week 40 (for 16-week treatment group); Week 48 (for 24-week treatment group)
Population: Standard population: The standard population includes all randomized participants who received at least one dose of study medication and who did not have any of the major protocol violations or deviations.
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 16 Weeks | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 24 Weeks
Number analyzed (Participants) | 679 | 630
percentage of participants | 65 | 76
Statistical Analysis 1: Comparison: PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 16 Weeks vs PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 24 Weeks; Test type: Non-Inferiority or Equivalence — These results indicated that sustained virological response achieved with 16 weeks of treatment was not equivalent to that achieved with 24 week of treatment; p < .0001, Cochran-Mantel-Haenszel; stratified by country and HCV genotype; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.46 to 0.76]

2. Secondary Outcome: Percentage of Participants With Virological Response at The End of Study Treatment
Description: Virological response was defined as the percentage of participants with undetectable HCV RNA at the completion of the study treatment. The negative assessment was required to be the last one collected in the Week 16 time window for the 16-week treatment group or in the Week 24 time window for the 24-week treatment group.
Time Frame: Week 16 (for 16-week treatment group); Week 24 (for 24-week treatment group)
Population: Standard population: The standard population included all randomized participants who received at least one dose of study medication and who did not have any of the major protocol violations or deviations.
Measure: Number; unit: Percentage of participants
Arm/Group | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 16 Weeks | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 24 Weeks
Number analyzed (Participants) | 679 | 630
Percentage of participants | 94 | 92
Statistical Analysis 1: Comparison: PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 16 Weeks vs PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 24 Weeks; Test type: Non-Inferiority or Equivalence — In the analysis based on the standard population, end of treatment virological response was equivalent in the two treatment arms (94% in the 16-week arm and 92% in the 24-week arm); p = 0.1941, Cochran-Mantel-Haenszel; stratified by country; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.86 to 2.03]

3. Secondary Outcome: Percentage of Participants Virological Response 12 Weeks Post-Treatment
Description: Virological response 12 weeks post-treatment was defined as the percentage of participants with undetectable HCV RNA 12 weeks after the completion of the study treatment . The negative assessment was required to be the last one collected in the week 28 time window for the 16- week treatment group or in the week 36 time window for the 24-week treatment group.
Time Frame: Week 28 (for 16-week treatment group); Week 36 (for 24-week treatment group)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 16 Weeks | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 24 Weeks
Number analyzed (Participants) | 679 | 630
Percentage of participants | 59 | 69
Statistical Analysis 1: Comparison: PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 16 Weeks vs PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 24 Weeks; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0003, Cochran-Mantel-Haenszel; stratified by country and HCV genotype; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.52 to 0.82]

4. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An adverse event was defined as any untoward medical occurrence that occurred during he course of the trial after study treatment had started. An adverse event was therefore any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug.
Time Frame: Up to Week 40 and Week 48
Population: Safety population: The safety population includes all randomized patients who received at least one dose of either study drug and had at least one post baseline safety assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 16 Weeks | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 24 Weeks
Number analyzed (Participants) | 731 | 728
Percentage of participants
  Any AE | 97 | 99
  Any SAE | 5 | 6

5. Secondary Outcome: Percentage of Participants With Marked Laboratory Abnormalities
Description: Participants with changes in Hematocrit: Fraction 0.36 - 0.60 g/dL, Hemoglobin: 11.0 -20.0 g/dL, WBC 3.0 - 18.0 g/dL, Platelets 100 - 700 g/dL, Basophils 0.00 - 0.30 g/dL, Lymphocytes 1.00 - 6.30 g/dL, Monocytes 0.08 - 2.00 g/dL, Neutrophils 1.50 or more g/dL, Eosinophils 0.00 - 1.50 g/dL , PTT 0 - 50 seconds, Alkaline Phosphatase 0 - 190 and ASAT 0 - 50 U/L, ALAT 0 - 60 U/L, Gamma - GT 0 - 120 U/L, Total Protein 55 - 87 g/L ;Albumin 27.0 or more g/L, Total Bilirubin 0 - 34.2 μmol/L, BUN 0 - 14.3 mmol/L, Creatinine 0 - 154 μmol/L, Free T3, T4 5 - 40 pmol/L, TSH 0.0 - 10.0 mU/L, Cholesterol 0.0 - 8.3 mmol/L; Triglycerides 0.00 - 2.83 mmol/L, Chloride 95 - 115 mmol/L; Potassium 3.0 - 6.0 mmol/L; Sodium 130 - 150 mmol/L, miscellaneous: Calcium 2.00 - 2.90 mmol/L; Phosphate 0.75 - 1.60 mmol/L; Blood Glucose (Random) 2.80 - 11.10 mmol/L, Uric Acid 0 - 600 μmol/L, Proteinuria, Glycosuria, Hematuria (Qualitative 0 to 4+) 0 - 1 were analysed for the laboratory abnormality.
Time Frame: Up to Week 40 and Week 48
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 16 Weeks | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 24 Weeks
Number analyzed (Participants) | 731 | 728
Percentage of participants
  Hematocrit (fraction)- low n=731,728 | 18 | 21
  Hemoglobin (g/dL)- low, n=731,727 | 15 | 16
  Platelets(10^9/L)- low,n=731,727 | 24 | 22
  Basophils(10^9/L)- high, n=731,727 | 0 | 0
  WBC (10^9/L)- low, n=731,727 | 64 | 71
  WBC (10^9/L)- high, n=731,727 | 0 | 0
  Eosinophils (10^9/L )- high, n=731,727 | 0 | 0
  Lymphocytes (10^9/L)- low, n=731,727 | 49 | 57
  Monocytes (10^9/L )- low, n=731,727 | 0 | 0
  Neutrophils (10^9/L)- low, n=731,727 | 69 | 75
  Partial throm.(seconds)- high, n=730,728 | 0 | 0
  Liver function: ALAT (SGPT) (U/L)- HIGH n=731,728 | 15 | 10
  Albumin (g/L)- low, n=730,728 | 0 | 0
  Alk. Phos.(U/L)- high,n=731,728 | 0 | 0
  ASAT (SGOT) (U/L)- high,n= 731,727 | 15 | 10
  GGT (U/L)- high,n=731,728 | 12 | 10
  Total bilirubin (umol/L)- high, n=731,728 | 0 | 0
  Total protein (g/L)- high, n=731,728 | 0 | 0
  Renal function: bun (mmol/L)- high, n=731,728 | 0 | 0
  Chloride (mmol/L)- high, n=731,728 | 0 | 0
  Chloride (mmol/L)- low, n=731,728 | 0 | 0
  Creatinine (umol/L)- high, n=731,728 | 0 | 0
  Potassium (mmol/L)- high, n=731,728 | 0 | 0
  Potassium (mmol/L)- low, n=731,728 | 0 | 0
  Sodium (mmol/L) - high, n=731,728 | 0 | 0
  Sodium (mmol/L)- low,n=731,728 | 0 | 0
  Thyroid function: free T4 (pmol/)- high, n=716,715 | 0 | 0
  Free T4 (pmol/L)- low, n=716,715 | 0 | 0
  TSH (mU/L)- high, n=716,715 | 2 | 6
  Miscellaneous: calcium (mmol/L)- low, n= 731,728 | 1 | 0
  Cholesterol (mmol/L)- high, n=730,728 | 0 | 0
  Phosphate (mmol/L)- high, n=730,728 | 2 | 2
  Phosphate (mmol/L)- low, n=730,728 | 18 | 21
  Random glucose (mmol/L)- high, n= 731,728 | 2 | 1
  Random glucose (mmol/L)- low, n= 731,728 | 2 | 0
  Triglycerides (mmol/L)- high, n=730,728 | 31 | 33
  Uric acid (umol/L)- high, n=730,728 | 2 | 2
  Urinalysis: glycosuria (0 to 4+)- high, n= 721,71 | 0 | 1
  Hematuria (0 to 4+) high, n= 721,716 | 4 | 4
  Proteinuria (0 to 4+) - high, n= 721,716 | 0 | 2

6. Secondary Outcome: Participants With Marked Abnormal Vital Signs
Description: Participants with changes in Systolic and diastolic blood pressure, heart rate were analysed abnormal vital signs.
Time Frame: Up to Week 40 and Week 48
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 16 Weeks | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 24 Weeks
Number analyzed (Participants) | 731 | 728
participants
  Diastolic BP, High, n=729,726 | 4 | 3
  Systolic BP, High, n=729,726 | 2 | 2
  Systolic BP, Low, n=729,726 | 9 | 2
  Heart Rate, High, n=728,725 | 2 | 3
  Heart Rate, Low, n=728,725 | 4 | 4

7. Secondary Outcome: Number of Participants With Highest Triglyceride Level
Description: Participants with triglyceride level above normal (i.e. < 200 mg/dL) were analysed.
Time Frame: Up to Week 40 and Week 48
Population: The safety population includes all randomized patients who received at least one dose of either study drug and had at least one post baseline safety assessment.
Measure: Number; unit: participants
Groups:
- PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 16 Weeks: Participants were administered 180 μg of PEG-IFN alfa-2a once weekly and 800 mg of ribavirin daily for 16 weeks.
Arm/Group | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 16 Weeks | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 24 Weeks
Number analyzed (Participants) | 731 | 728
participants
  200 - 400 mg/dL | 280 | 284
  >400 - 1000 mg/dL | 117 | 138
  >1000 mg/dL | 17 | 14

ADVERSE EVENTS:
Time Frame: Up to week 48
Description: An adverse event was defined as any untoward medical occurrence that occurred during the course of the trial after study treatment had started. An adverse event was therefore any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug.
Arm/Group | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 16 Weeks | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 24 Weeks
Serious Adverse Events (participants affected / at risk) | 34/731 | 47/728
Other Adverse Events (participants affected / at risk) | 696/731 | 713/728
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 16 Weeks (N=731) | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 24 Weeks (N=728)
Pneumonia (Infections and infestations) | 3 | 3
Cellulitis (Infections and infestations) | 2 | 0
Diverticulitis (Infections and infestations) | 0 | 2
Pyelonephritis (Infections and infestations) | 2 | 0
Staphylococcal infection (Infections and infestations) | 2 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 1
Abscess limb (Infections and infestations) | 1 | 0
Chronic tonsillitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Keratitis herpetic (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Meningitis viral (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Appendicitis perforated (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Volvulus of bowel (Gastrointestinal disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 4
Depression (Psychiatric disorders) | 0 | 2
Drug dependence (Psychiatric disorders) | 0 | 1
Homicidal ideation (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 2
Overdose (Injury, poisoning and procedural complications) | 1 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebra injury (Injury, poisoning and procedural complications) | 0 | 1
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Mononeuropathy multiplex (Nervous system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 1 | 0
Retinal artery thrombosis (Eye disorders) | 1 | 0
Retinal exudates (Eye disorders) | 0 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 16 Weeks (N=731) | PEG-IFN Alfa-2a 180μg + Ribavirin 800 mg 24 Weeks (N=728)
Vision blurred (Eye disorders) | 37 | 38
Abdominal pain (Gastrointestinal disorders) | 36 | 47
Abdominal pain upper (Gastrointestinal disorders) | 43 | 40
Diarrhoea (Gastrointestinal disorders) | 123 | 165
Dry mouth (Gastrointestinal disorders) | 27 | 37
Dyspepsia (Gastrointestinal disorders) | 33 | 42
Nausea (Gastrointestinal disorders) | 230 | 247
Vomiting (Gastrointestinal disorders) | 87 | 78
Asthenia (General disorders) | 95 | 108
Chills (General disorders) | 150 | 146
Fatigue (General disorders) | 356 | 393
Injection site erythema (General disorders) | 79 | 103
Pain (General disorders) | 61 | 73
Pyrexia (General disorders) | 187 | 184
Upper respiratory tract infection (Infections and infestations) | 26 | 39
Anorexia (Metabolism and nutrition disorders) | 74 | 74
Decreased appetite (Metabolism and nutrition disorders) | 69 | 71
Arthralgia (Musculoskeletal and connective tissue disorders) | 139 | 152
Back pain (Musculoskeletal and connective tissue disorders) | 69 | 68
Myalgia (Musculoskeletal and connective tissue disorders) | 188 | 199
Pain in extremity (Musculoskeletal and connective tissue disorders) | 30 | 39
Disturbance in attention (Nervous system disorders) | 39 | 54
Dizziness (Nervous system disorders) | 76 | 91
Headache (Nervous system disorders) | 285 | 337
Anxiety (Psychiatric disorders) | 78 | 80
Depression (Psychiatric disorders) | 148 | 163
Insomnia (Psychiatric disorders) | 234 | 272
Irritability (Psychiatric disorders) | 156 | 184
Cough (Respiratory, thoracic and mediastinal disorders) | 88 | 87
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 88 | 93
Alopecia (Skin and subcutaneous tissue disorders) | 86 | 102
Dry skin (Skin and subcutaneous tissue disorders) | 63 | 86
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 37 | 47
Pruritus (Skin and subcutaneous tissue disorders) | 107 | 140
Rash (Skin and subcutaneous tissue disorders) | 124 | 118

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.